CLINICAL TRIAL: NCT04387331
Title: The Postoperative Head Position as a Predictor of the Surgical Outcome After DMEK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peter Wiedemann (Other)
Collaborators: Institut für Angewandte Trainingswissenschaft (Unknown)
Responsible Party: Sponsor-Investigator, Peter Wiedemann, Director, University of Leipzig
Organization: University of Leipzig (Other)
Other Study IDs: 287/19-ek
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; Pseudophakic Bullous Keratopathy; Chemical Burn of Cornea; Posterior Polymorphous Corneal Dystrophy
Keywords: Descemet Membrane Endothelial Keratoplasty; DMEK; Fuchs Endothelial Corneal Dystrophy; Pseudophakic Bullous Keratopathy; Chemical Burn of Cornea; Posterior Polymorphous Corneal Dystrophy; Postoperative Head Position; Corneal Transplantation; Head Tracking Sensor
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Dystrophy, Posterior Polymorphous, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the influence of postoperative head position on clinical outcomes after DMEK via a wearable sensor.

DETAILED DESCRIPTION:
After Descemet Membrane Endothelial Keratoplasty (DMEK) patients are recommended to keep a strict supine position within the first few days after surgery in order to attach the graft to the corneal stroma. It has not yet been investigated to what extent the head position actually has an effect on the outcome.

In this study, the participants head position will be continuously monitored within the first three days after DMEK. Participants wear a headband in which a small sensor is inserted. The degree of deviation from the neutral position will then be correlated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing DMEK

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Descemet Membrane Endothelial Keratoplasty during the study are offered to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Corneal Endothelial Cell Density | three months after surgery
  measured in cells/mm2

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | prior to surgery, three and six months after surgery
  measured in logMAR
Central Corneal Thickness | prior to surgery, three and six months after surgery
  measured in μm
Number of Re-Bubblings | six months after surgery
  need of surgical intervention after DMEK in order to attach the graft
Corneal Endothelial Density | six months after surgery
  measured in cells/mm"

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wiedemann, MD, Study Director — University of Leipzig
Locations (1):
- Leipzig University Hospital, Department of Ophthalmology, Leipzig, Saxony, Germany